CLINICAL TRIAL: NCT02569203
Title: Effects of Enteral Formula Including Immune-modulating Nutrients on Clinical Course and Immune Function in Critically Ill Patients
Brief Title: Effect of Immune-enhancing Enteral Nutrition on Immunomodulation in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: BT_ICU_immune
Record Dates: First submitted 2015-09-24; First posted 2015-10-06 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- control group (Placebo Comparator): standard enteral nutrition
  Interventions: Dietary Supplement: standard enteral nutrition
- test group I (Experimental): high-protein enteral nutrition of immune modulating nutrients enriched with β-glucan
  Interventions: Dietary Supplement: high-protein enteral nutrition of immune modulating nutrients enriched with β-glucan
- test group II (Experimental): high-protein enteral nutrition of immune modulating nutrients without β-glucan
  Interventions: Dietary Supplement: high-protein enteral nutrition of immune modulating nutrients without β-glucan

INTERVENTIONS:
Dietary Supplement: standard enteral nutrition — standard enteral nutrition
  Other Names: control group
  Arms: control group
Dietary Supplement: high-protein enteral nutrition of immune modulating nutrients enriched with β-glucan — high-protein enteral nutrition of immune modulating nutrients enriched with β-glucan
  Other Names: test group I
  Arms: test group I
Dietary Supplement: high-protein enteral nutrition of immune modulating nutrients without β-glucan — high-protein enteral nutrition of immune modulating nutrients without β-glucan
  Other Names: test group II
  Arms: test group II

SUMMARY:
To determine whether high-protein (24% of total calorie from protein) enteral nutrition of immune modulating nutrients (eg, ω-3 fatty acids and antioxidants) enriched with β-glucan stimulates immune functions compared with standard enteral nutrition (control: 20% of total calorie from protein) or high-protein (24% of total calorie from protein) enteral nutrition of immune modulating nutrients without β-glucan in critically ill patients.

DETAILED DESCRIPTION:
To determine whether high-protein (24% of total calorie from protein) enteral nutrition of immune modulating nutrients (eg, ω-3 fatty acids and antioxidants) enriched with β-glucan stimulates immune functions compared with standard enteral nutrition (control: 20% of total calorie from protein) or high-protein (24% of total calorie from protein) enteral nutrition of immune modulating nutrients without β-glucan in critically ill patients. In a randomized double-blind placebo-controlled study, 30 patients consumed 1 of 3 enteral nutrition: control, enteral nutrition of immune modulating nutrients enriched with β-glucan (250mg/L) or enteral nutrition of immune modulating nutrients without β-glucan. Enteral nutrition was initiated within 24 hours of ICU admission and continued during the ICU stay for a 7 days.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients

Exclusion Criteria:

* ICU patients who could not receiving enteral nutrition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline NK cell activity at 7 days | at baseline and 7 days follow-up
  NK cell activity (%)

SECONDARY OUTCOMES:
Change from baseline IL-12 at 7 days | at baseline and 7 days follow-up
  IL-12 (pg/mL)
Change from baseline hs-CRP at 7 days | at baseline and 7 days follow-up
  hs-CRP (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Lee, Ph. D., Principal Investigator — Dept. of Food and Nutrition, College of Human Ecology, Yonsei University, 50 Yonsei-ro, Seodaemun-gu, Seoul, 120-749, South Korea

REFERENCES:
- [Derived] Lee JG, Kim YS, Lee YJ, Ahn HY, Kim M, Kim M, Cho MJ, Cho Y, Lee JH. Effect of Immune-Enhancing Enteral Nutrition Enriched with or without Beta-Glucan on Immunomodulation in Critically Ill Patients. Nutrients. 2016 Jun 2;8(6):336. doi: 10.3390/nu8060336. PMID 27271657